CLINICAL TRIAL: NCT04613921
Title: Liver Transplantation in Patients With CirrHosis and Severe Acute-on-Chronic Liver Failure (ACLF): iNdications and outComEs
Brief Title: Liver Transplantation in Patients With CirrHosis and Severe Acute-on-Chronic Liver Failure: iNdications and outComEs
Acronym: CHANCE
Status: Recruiting | Type: Observational
Sponsor: European Foundation for Study of Chronic Liver Failure (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/01325
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Liver Diseases; Liver Cirrhosis; Acute-On-Chronic Liver Failure; Liver Transplant; Complications
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA and RNA Description: peripherical serum, plasma, urine, saliva, liver biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: patients listed for liver transplantation with ACLF-2 or 3 at the time of listing or developing ACLF 2-3 while on the waiting list (n=2,000)
  Interventions: Other: Observational Protocol
- Group 2: patients listed for liver transplantation with decompensated cirrhosis without ACLF-2 or 3 and poor liver function (MELD > 20) at the time of listing (n=500)
  Interventions: Other: Observational Protocol
- Group 3: patients having ACLF-2 or 3, are assessed for inclusion in the waiting list, but are finally not listed for liver transplantation (n=500)
  Interventions: Other: Observational Protocol

INTERVENTIONS:
Other: Observational Protocol — The cohorts will be followed for one year after LT transplantation except for group 3 (1-year follow-up after inclusion)

SUMMARY:
Management of ACLF is mainly supportive. The poor outcomes lead physicians to consider liver transplantation as an option, even if controversial. In sicker recipients, LT results in immediate survival, but poor medium-term survival rates in some studies. The scarcity of deceased donors obliges to maximize LT success. Alternative strategies, as living-donor LT, should be explored. LDLT has impressive results in Eastern centers, but it is restrained in Western countries, due to potential life-threatening complications in the donor.

DETAILED DESCRIPTION:
The aim of this study is to compare 1-year graft and patient survival rates after liver transplantation (LT) in patients with ACLF-2 or 3 at the time of LT, with patients with decompensated cirrhosis without ACLF-2 or 3 at the time of LT and also with transplant-free survival of patients with ACLF-2 or 3 not listed for LT.

Secondary objectives are as follows:

* To assess the proportion of patients with ACLF-2 or 3 referred to transplant team who are listed or not and reasons of this decision.
* To evaluate the outcomes of patients listed with ACLF-2 or 3 on the waiting list compared with those of patients listed with decompensated cirrhosis without ACLF-2 or 3.
* To define independent predictive factors of death/delisting on the waiting list for patients listed with ACLF-2 or 3 and develop a new prognostic model based on ACLF criteria to predict mortality on the waiting list and to improve the allocation of organs.
* To compare the characteristics of accepted grafts for patients listed with ACLF-2 or 3 with those of patients listed with decompensated cirrhosis without ACLF-2 or 3 and their impact on post-LT outcomes.
* To explore independent predictive factors of death after LT for patients transplanted with ACLF-2 or 3 to design futility criteria for LT.
* To compare post-LT survival rates of patients with ACLF-2 or 3 at listing and patients without ACLF at listing who develop ACLF-2 or 3 on the waiting list.
* To compare post-LT quality of life (QoL) for patients listed with ACLF-2 or 3 with those of patients listed with decompensated cirrhosis without ACLF-2 or 3.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subject ≥18 years of age.

  2. Subjects with diagnosis of liver cirrhosis (based on clinical, laboratory, endoscopic, and ultrasonographic features or on histology).

  3. Subjects who have been hospitalized for acute decompensation of liver cirrhosis and referred to the transplant team:
* Group 1: patients listed for liver transplantation with ACLF-2 or 3 at the time of listing or developing ACLF 2-3 while on the waiting list.
* Group 2: patients listed for liver transplantation with decompensated cirrhosis without ACLF-2 or 3 and poor liver function (MELD>20) at the time of listing.
* Group 3: patients having ACLF-2 or 3, are assessed for inclusion in the waiting list, but are finally not listed for liver transplantation.

  4. Patients (or trusted person, family member or close relation if the patient is unable to express consent) who have been informed and signed their informed consent Inclusion criteria

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute or subacute liver failure. Patients with hepatocellular carcinoma Subjects listed for transplantation other than liver or liver-kidney transplant.
  Subjects with previous liver transplantation. Vulnerable population. Pregnant and/or breastfeeding woman Patients with relevant comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  survival

CONTACTS AND LOCATIONS:
Locations (106):
- United States (18):
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine (Scott & White), Dallas, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Baylor St. Luke's Medical Centre, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
- Argentina (3):
  - Austral University Hospital, Buenos Aires
  - Hospital Alemán, Buenos Aires
  - Italian Hospital in Buenos Aires, Buenos Aires
- Australia (3):
  - Austin Hospital, Heidelberg
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal Prince Alfred Hospital, Sydney
- Medical University of Vienna, Department of Transplant Surgery, Vienna, Austria
- Belgium (3):
  - CUB Erasme Hospital, Brussels
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven
- Brazil (3):
  - Walter Cantídio University Hospital, Fortaleza
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital das Clínicas da Universidade de São Paulo, São Paulo
- Canada (2):
  - University of Alberta, Edmonton
  - University of Toronto, Multiorgan Transplant Program, Toronto
- Pablo Tobón Uribe Hospital, Medellín, Colombia
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- France (9):
  - APHP Beaujon, Clichy
  - APHP Henri Mondor, Créteil
  - Hôpital de la Croix-Rousse, Lyon
  - CHU Montpellier-Hôpital Saint Eloi, Montpellier
  - APHP Hôpitaux Universitaires Pitié Salpêtrière, Paris
  - CHU Rennes, Hôpital De Pontchaillou, Rennes
  - Hautepièrre Hospital, Service de Réanimation Médicale, Strasbourg
  - Trousseau Hospital,, Tours
  - Hôpital Paul Brousse, Villejuif
- Germany (15):
  - University Hospital Regensburg, Regensburg, Eastern Bavaria
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel, Schleswig-Holstein
  - University Hospital Aachen, Aachen
  - Charité University Hospital, Berlin
  - Goethe University Clinic, Frankfurt
  - University Medical Center, Hamburg Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Heidelberg, Heidelberg
  - Jena University Hospital, Jena
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel
  - Leipzig University Hospital, Leipzig
  - University Hospital Mainz, Mainz
  - LMU Großhadern, Munich
  - UKM Muenster, Münster
  - University Hospital Tübingen, Tübingen
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- India (12):
  - Aster CMI Hospital, Bengaluru, Karnataka
  - Kasturba Hospital, Mumbai, Maharashtra
  - Seth GSMC & KEM Hospital, Mumbai, Maharashtra
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Mahatma Gandhi University of Medical Sciences and Technology, Jaipur, Rajasthan
  - Dr.Rela Institute & Medical Centre, Chennai
  - Fortis Hospital Noida, FEHI, FMRI, Gurugramam
  - Medanta Medicity, Gurugramam
  - Amrita Institute of Medical Sciences, Kochi
  - Global Hospital. Super speciality & transplant centre, Mumbai
  - Max Saket Hospital, New Delhi
  - Yashoda Hospitals, Secunderabad
- Italy (5):
  - Ospedale Papa Giovanni XXIII-, Bergamo
  - S.Orsola Hospital - Alma Mater Studiorum University of Bologna, Bologna
  - Ca' Granda. Policlinico Milano, Milan
  - Niguarda Hospital, Milan
  - University and Hospital of Padova, Padua
- Japan (5):
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Tokyo University Hospital, Tokyo
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico
- Netherlands (2):
  - University Medical Center Groningen (UMCG), Groningen
  - Erasmus MC University Medical Center, Rotterdam
- Auckland City Hospital- New Zealand Liver Transplant Unit, Auckland, New Zealand
- Medical University of Warsaw, Dept. of General, Transplant & Liver Surgery, Warsaw, Poland
- Hospital Curry Cabral, Lisbon, Portugal
- Samsung Medical Center, Seoul, South Korea
- Spain (7):
  - Hospital Clinic in Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Karolinska Institutet, Stockholm, Stockholm County, Sweden
- Geneva University Hospital (HUG), Geneva, Switzerland
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan
- Turkey (Türkiye) (2):
  - Inonu University, Liver Transplantation Institute, Malatya, Anatolia
  - Istanbul Memorial Bahcelievler Hospital, Istanbul
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Scottish Liver Transplant Unit, Royal Infirmary, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - King's College Hospital, London
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustot T, Fernandez J, Garcia E, Morando F, Caraceni P, Alessandria C, Laleman W, Trebicka J, Elkrief L, Hopf C, Solis-Munoz P, Saliba F, Zeuzem S, Albillos A, Benten D, Montero-Alvarez JL, Chivas MT, Concepcion M, Cordoba J, McCormick A, Stauber R, Vogel W, de Gottardi A, Welzel TM, Domenicali M, Risso A, Wendon J, Deulofeu C, Angeli P, Durand F, Pavesi M, Gerbes A, Jalan R, Moreau R, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Clinical Course of acute-on-chronic liver failure syndrome and effects on prognosis. Hepatology. 2015 Jul;62(1):243-52. doi: 10.1002/hep.27849. Epub 2015 May 29. PMID 25877702
- [Background] Artru F, Louvet A, Ruiz I, Levesque E, Labreuche J, Ursic-Bedoya J, Lassailly G, Dharancy S, Boleslawski E, Lebuffe G, Kipnis E, Ichai P, Coilly A, De Martin E, Antonini TM, Vibert E, Jaber S, Herrerro A, Samuel D, Duhamel A, Pageaux GP, Mathurin P, Saliba F. Liver transplantation in the most severely ill cirrhotic patients: A multicenter study in acute-on-chronic liver failure grade 3. J Hepatol. 2017 Oct;67(4):708-715. doi: 10.1016/j.jhep.2017.06.009. Epub 2017 Jun 21. PMID 28645736
- [Background] Sundaram V, Jalan R, Wu T, Volk ML, Asrani SK, Klein AS, Wong RJ. Factors Associated with Survival of Patients With Severe Acute-On-Chronic Liver Failure Before and After Liver Transplantation. Gastroenterology. 2019 Apr;156(5):1381-1391.e3. doi: 10.1053/j.gastro.2018.12.007. Epub 2018 Dec 18. PMID 30576643